CLINICAL TRIAL: NCT06701422
Title: Targeting Cervical Epidural Spinal Cord Stimulation for Functional Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason Carmel, Associate Professor, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AAAV1303; CDMRP-SC230233 (Other Grant/Funding Number: U.S. Department of Defense, Congressionally Directed Medical Research Programs (CDMRP))
Record Dates: First submitted 2024-11-13; First posted 2024-11-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cervical Spinal Cord Injury; Tetraplegia/Tetraparesis; Cervical Myelopathy
Keywords: spinal cord injury; upper-limb muscle activation; cervical spinal cord; myelopathy
MeSH Terms: conditions — Quadriplegia; Spinal Cord Injuries; Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 - Intraoperative Participants (Experimental): Motor evoked responses responses (MEPs) to epidural electrical stimulation (EES) will be tested at cervical segments with and without myelopathy in participants with cervical myelopathy.
  Interventions: Procedure: Intraoperative stimulation of the cervical spinal cord

INTERVENTIONS:
Procedure: Intraoperative stimulation of the cervical spinal cord — The surgeon will place spinal cord electrodes on the epidural surface, with stimulation sites identified using preoperative MRI. Recruitment curves will be generated by systematically increasing the stimulation intensity across various parameter combinations, including frequency, pulse count, pulse shape, and electrode-specific properties such as size, separation, and arrangement.

SUMMARY:
The proposed study seeks to understand how the cervical spinal cord should be stimulated after injury through short-term physiology experiments that will inform a preclinical efficacy trial. The purpose of this study is to determine which cervical levels epidural electrical stimulation (EES) should target to recruit arm and hand muscles effectively and selectively in spinal cord injury (SCI).

DETAILED DESCRIPTION:
For people with cervical spinal cord injury (SCI), regaining hand and arm function is their highest priority. Epidural stimulation enables recovery of walking and autonomic function in people with chronic SCI, but how the spinal cord should be stimulated to restore arm and hand function is not known. This project seeks to advance our understanding of how best to apply epidural electrical stimulation (EES) after cervical SCI using complementary experiments in humans and rats. This improved understanding will be used to conduct a preclinical study of the efficacy of different sites of cervical spinal cord stimulation.

ELIGIBILITY:
Inclusion Criteria:

•Clinical indication for cervical spine surgery.

Exclusion criteria:

•Stimulation devices in the neck or chest (e.g., vagal nerve stimulation, cardiac patients with pacemakers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of epidural SCS | 0-100 milliseconds after each stimulation event during the experiment
  Efficacy of stimulation is calculated as 1/threshold for provoking an motor evoked potentials. The threshold will be calculated from the recruitment curves.
Selectivity of epidural SCS | 0-100 milliseconds after each stimulation event during the experiment
  Selectivity is calculated from the recruitment curves of the target muscle compared to non-targeted muscles.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - The Daniel and Jane Och Spine Hospital at NewYork-Presbyterian/Allen, New York, New York

IPD SHARING:
Plan to Share IPD: No